CLINICAL TRIAL: NCT00856414
Title: Patient Satisfaction With Treatment of BOTOX® Cosmetic for the Temporary Correction of Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BTX-0806
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Results first posted 2011-12-12 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Skin Aging
MeSH Terms: interventions — Botulinum Toxins, Type A

ARMS (1):
- 1 (Experimental): botulinum toxin Type A 20U
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — 20U, up to two injections administered intramuscularly into the glabella (2 in each side of the corrugators and 1 in the procerus)
  Other Names: BOTOX®

SUMMARY:
This study evaluates the patient satisfaction and onset of effect following treatment with botulinum toxin Type A in the treatment of glabellar rhytids (frown lines)

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of any race, 35-55 years of age
* Moderate to severe glabellar wrinkles (lines between the eyebrows)

Exclusion Criteria:

* Previous botulinum toxin therapy
* Subjects who are pregnant, breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control
* Subjects planning a facial cosmetic procedure or visible scars
* Previous cosmetic surgery to the upper face
* Medical condition that may increase their risk of exposure to botulinum toxin including diagnosed Myasthenia Gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis, or any other disease that might interfere with neuromuscular function
* History of facial nerve palsy
* Allergy or sensitivity to any component of the study medication

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2009-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- United States (2):
  - West Palm Beach, Florida
  - Livonia, Michigan

REFERENCES:
- [Background] Beer KR, Boyd C, Patel RK, Bowen B, James SP, Brin MF. Rapid onset of response and patient-reported outcomes after onabotulinumtoxinA treatment of moderate-to-severe glabellar lines. J Drugs Dermatol. 2011 Jan;10(1):39-44. PMID 21197522

RESULTS

PARTICIPANT FLOW:
Groups:
- Botulinum Toxin Type A 20U: botulinum toxin Type A 20U
Period: Overall Study
Arm/Group | Botulinum Toxin Type A 20U
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Botulinum Toxin Type A 20U
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 43.5 [35.1 to 56.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: The First Visit Onset of Efficacy as Measured by Physician Assessment
Description: The first visit onset of efficacy as measured by physician assessment. Onset is determined by a yes/no answer to the question "Since injecting the patient, have you noticed any effect on the appearance of the patient's frown lines (lines between the eyebrows)?" at days 2, 3, 4, 7, and 14.
Time Frame: 14 Days
Population: Intent to Treat defined as all patients who started the study
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Botulinum Toxin Type A 20U
Number analyzed (Participants) | 45
Number of Days | 2.2 (0.55)

2. Primary Outcome: The First Visit Onset of Efficacy as Measured by Subject Assessment
Description: The first visit onset of efficacy as measured by subject assessment. Onset is determined by a yes/no answer to the question "Since being injected, have you noticed any effect on the appearance of your frown lines (lines between the eyebrows)?" at days 2, 3, 4, 7, and 14.
Time Frame: 14 Days
Population: Intent to Treat defined as all patients who started the study
Measure: Mean (Standard Deviation); unit: Number of Days
Arm/Group | Botulinum Toxin Type A 20U
Number analyzed (Participants) | 45
Number of Days | 1.84 (1.01)

3. Secondary Outcome: Average Subject Assessment Score in Improvement of Appearance of Frown Lines
Description: Average subject assessment score in improvement of appearance of frown lines (lines between the eyebrows) as measured by a 7-point scale (1=very much improved and 7=very much worse)on a daily basis. The average scores over the 1st diary week (1-7 days) and the 2nd diary week (8-14 days) are presented.
Time Frame: 14 Days
Population: Intent to Treat defined as all patients who started the study
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 20U
Number analyzed (Participants) | 45
Scores on a Scale
  1st Diary Week | 1.73 (0.65)
  2nd Diary Week | 2.64 (0.57)

4. Secondary Outcome: Change From Baseline in Patient Satisfaction as Measured by Facial Line Outcome (FLO) Questionnaire Score
Description: Change from baseline in patient satisfaction as measured by FLO questionnaire comprised of 11 items that assess subject's perceptions about specific aspects of their facial lines for the previous 7 days. Each question is scored on a 11-point scale (0=not at all, 5=somewhat, 10=very much) and the sums are converted to the total FLO score. The minimum total FLO score is 0 (worst) and the maximum total FLO score is 100 (best). The total FLO score was calculated at baseline and Day 14. A positive number change from baseline indicates an improvement.
Time Frame: Baseline, Day 14
Population: Intent to Treat defined as all patients who started the study
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Botulinum Toxin Type A 20U
Number analyzed (Participants) | 45
Scores on a Scale
  Baseline | 32.97 (19.91)
  Change from Baseline at Day 14 | 38.55 (28.20)

5. Secondary Outcome: Percentage of Patients Reporting Self-Perception of Age (SPA)
Description: Percentage of patients reporting their SPA. SPA is measured by a questionnaire. Patients were asked to compare their facial appearance to their current age. Response options were "Looking younger", "Looking current age", and "Looking older". Results for each response are presented for Baseline and Day 14.
Time Frame: Baseline, Day 14
Population: Intent to Treat defined as all patients who started the study
Measure: Number; unit: Percentage of patients
Arm/Group | Botulinum Toxin Type A 20U
Number analyzed (Participants) | 45
Percentage of patients
  Baseline Looking Younger | 22.2
  Baseline Looking Current Age | 40.0
  Baseline Looking Older | 37.8
  Day 14 Looking Younger | 42.2
  Day 14 Looking Current Age | 44.4
  Day 14 Looking Older | 13.3

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin Type A 20U
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo